CLINICAL TRIAL: NCT06688955
Title: Evaluation of the Microbiological and Organizational Impact of the Use of Bacteriologically Controlled Water in COLOscopy for an Evolution of Our Practices Towards a More Ecoresponsible Endoscopic Activity COLO SOUS L'EAU
Brief Title: Microbiological and Organizational Impact of the Use of Bacteriologically Controlled Water in COLOscopy
Acronym: COLOSOUS L'EAU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2023/38
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Colonoscopy
Keywords: COLONOSCOPY; WATER; microbiological safety; organization; ecological impacT; plastic waste
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with Bacteriologically Controlled Water procedure (Experimental): patient with colonoscopy with Bacteriologically Controlled Water procedure
  Interventions: Procedure: Colonoscopy with Bacteriological Controlled Water

INTERVENTIONS:
Procedure: Colonoscopy with Bacteriological Controlled Water — Patient with coloscopy which used Bacteriological Controlled Water : Collection of 250 ml of bacteriologically controlled water from the wash bottle at the end of each water-assisted colonoscopy to test for enterobacteria and fecal streptococci

SUMMARY:
A joint opinion of the SFED and the SF2H recommends to orient our colonoscopy practices towards the use of bacteriologically controlled water in reusable bottles for colonic irrigation. To date, no study exists to validate the proposed set-up. Our main objective is therefore to evaluate the microbiological safety of the use of bacteriologically controlled water, in particular the absence of retro contamination of the water in the wash bottle by the faecal flora of the patient undergoing colonoscopy, in order to be able to generalise this practice

DETAILED DESCRIPTION:
Colonoscopy is the reference examination for colon exploration. Since 2021, international recommendations recommend the practice of "water-exchange" which consists in performing colonoscopies by irrigating the colon with water, continuously and without insufflation. This technique facilitates the progression of the colonoscope, reduces pain and the risk of perforation for the patient, and improves the detection and resection of polyps. However, it requires a large volume of water, about 1L per patient. We currently use sterile water in single-use bottles. In order to propose a way to limit the production of waste in endoscopy, the SFED and the SF2H have published an opinion proposing to orient our practice towards the use of EBM packaged in reusable bottles. To date, no study has validated the set-up proposed in this advice. We therefore propose to ensure the microbiological safety of the use of EBM during water-assisted colonoscopies before generalizing this practice. A microbiological sample of 200 ml of EBM contained in the wash bottle at the end of each colonoscopy will be collected for bacteriological analysis. In addition, the use of reusable bottles requires the implementation of a maintenance and reconditioning circuit, and therefore a reorganization within the technical platform, the feasibility and acceptability of which must be evaluated by the professionals. Finally, we will also evaluate the carbon footprint of the sterilization circuit and compare the weight of waste related to the current practice, sterile water versus the use of EBM. This study would be the pilot phase for a larger study on the ecological and medico-economic impact of the use of bacteriologically controlled water in endoscopy

ELIGIBILITY:
Inclusion Criteria:

* All patients with a colonoscopy indication whose examination is scheduled in room 4, on a Monday and Tuesday shift (8:30 a.m. - 1:30 p.m.)
* Male or female of legal age at the time the colonoscopy is ordered
* Patient willing to participate in the study
* Person affiliated with or benefiting from a social security plan

Exclusion Criteria:

* Pregnant woman
* Patient of legal age under guardianship or protected person
* Patient requiring indigo-carmine chromoendoscopy
* Patient requiring an emergency colonoscopy
* Patient not affiliated to the social security system

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of back contamination | inclusion visit
  Rate of back contamination after colonoscopy using the EBM procedure. The absence of retro-contamination is defined as the absence of fecal flora (enterobacteria and fecal streptococci) in the wash bottle during the bacteriological analysis of the EBM microbiological samples taken after each colonoscopy

SECONDARY OUTCOMES:
Workload | Inclusion visit
  Estimation of the workload in minutes, per person involved and for each phase of the reusable vial circuit
Satisfaction and acceptability healthcare professionals | Inclusion visit
  Evaluation of satisfaction and acceptability among healthcare professionals using the French version of the System Usability Scale (FSUS).
Acceptability patient | Inclusion visit
  Assessment of patient acceptability of Bacteriologically Controlled Water use by counting the total number of patients offered the study to obtain 40 consents
Infectious episode | DAY 1 VISIT AND DAY 7 VISIT
  Monitoring the occurrence of an infectious episode (D+1 and D+7) characterized by the occurrence of a fever episode higher than 38.5°C.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur BERGER, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux - Hôpital haut Lévêque, Pessac, France